CLINICAL TRIAL: NCT06315452
Title: FREQUENCY OF VITAMIN D DEFICIENCY IN PREMATURE NEWBORN BORN BEFORE 32 WEEKS AND/OR WITH A BIRTH WEIGHT UNDER 1500g
Acronym: PremaVitaD
Status: Active, not recruiting | Type: Observational
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Other Study IDs: PremaVitaD
Record Dates: First submitted 2024-03-11; First posted 2024-03-18 (Actual); Last update posted 2024-03-18 (Actual); Status verified 2024-03

CONDITIONS: Vitamin D Deficiency
MeSH Terms: conditions — Vitamin D Deficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Vitamin D plays an important role in phosphocalcic metabolism and bone homeostasis in newborns. Premature newborns are at risk of vitamin D deficiency and may require supplementation. In this context, the French Society of Pediatrics (Société Française de Pédiatrie) recommends systematic vitamin D testing at 1 month.

The aim of this study was to determine the frequency of vitamin D deficiency in premature newborns.

ELIGIBILITY:
Inclusion Criteria:

* Premature newborns born at a gestational age less than 32 weeks and/or birth weight less than 1500g
* Having received at least one dosage of 25 OH vitamin D.-

Exclusion Criteria:

* - Newborn whose parents or legal guardian refuse the use of their data for this research

Ages: 1 Day to 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: PREMATURE NEWBORN BORN BEFORE 32 WEEKS AND/OR WITH A BIRTH WEIGHT UNDER 1500g
Sampling Method: Non-Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2024-02-01 (Actual); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
Vitamine D deficiency frequency | 6 months
  25-OH Vitamine D values will be collected for premature newborn , born before 32 weeks, or with a birth weight under 1500g.
  A 25-OH Vitamine D blood value under 20µg/L is considered as a vitamine D deficiency

SECONDARY OUTCOMES:
vitamine D deficiency and maternal or feotal caracteristics | 6months
  correlation between vitamine D deficiency and maternal or feotal caracteristics
vitamine D deficiency and premature newborn comorbidities | 6 months
  correlation between vitamine D deficiency and premature newborn comorbidities
effect of supplementation | 6months
  Number (proportion) of children with normalized 25 OH vitamin D levels after Vitamine D supplementation according to neonatal department protocol.

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Saint Joseph, Paris, France